CLINICAL TRIAL: NCT04324918
Title: Efficacy and Safety of HCP1102 in Patients With Perennial Allergic Rhinitis : A Randomized, Double-blind, Active-controlled, Multicenter Phase 3 Clinical Trial
Brief Title: Efficacy and Safety of HCP1102 Capsule in Patients With Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-MOLZ-303
Record Dates: First submitted 2020-02-04; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HCP1102 (Experimental)
  Interventions: Drug: HCP1102
- HGP1408 (Active Comparator)
  Interventions: Drug: HGP1408

INTERVENTIONS:
Drug: HCP1102 — The participants will receive tretment of HCP1102(combination of Montelukast + Levocetrizine), orally, once daily for 4weeks.
  Arms: HCP1102
Drug: HGP1408 — The participants will receive tretment of HGP1408(Levocetrizine), orally, once daily for 4weeks.
  Arms: HGP1408

SUMMARY:
Efficacy and safety of HCP1102 in patients with perennial allergic rhinitis :

A randomized, double-blind, active-controlled, multicenter phase 3 clinical trial

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least 2 years history of PAR prior to the study
* Positive results of skin prick test
* Patients who provided a signed written informed consent form
* Patients who are able and willing to complete subject diaries
* Patients who agree to maintain consistency in their surroundings throughout the study period

Exclusion Criteria:

* Patients also with non-allergic rhinitis with different causes.
* Patients with severe asthma.
* History of acute • chronic sinusitis within 1 month of Visit 1
* History of intranasal surgeries within 3 months of Visit 1
* Initiation of immunotherapy or dose modification within 1 month prior to Visit 1
* Upper respiratory infections including cold and systemic infections within 3 weeks of Visit 1.
* Chronic use of tricyclic antidepressants, beta agonists, bronchodilators, etc. that may affect the efficacy of study drug.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Change of Mean Daytime Nasal Symptom Score | base line, 3-4week(2weeks)
  Daytime nasal symptoms included rhinorrhea, nasal obstruction, sneezing, and itching, each scored from 0 to 3 (0 = none, 1 = mild, 2 = moderate and 3 = severe).

SECONDARY OUTCOMES:
Change of Mean Nighttime Nasal Symptom Score | baseline, 3-4week(2weeks)
  Nighttime nasal symptoms included nasal obstruction awakening (0 = none; 1 = mild; 2 = moderate; 3 = severe), difficulty getting to sleep (0 = not at all; 1 = little; 2 = moderate; 3 = severe), and nighttime awakening (0 = not at all; 1 = once; 2 = more than once; 3 = awake all night).

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Su Kim, M.D., Ph.D., Principal Investigator — Gangnam Severance Hospital
Locations (1):
- Gangnam Severance Hospital., Seoul, South Korea